CLINICAL TRIAL: NCT04123106
Title: Bilateral Erector Spinae Plane Block (ESP Block) Versus Local Anesthetic (LA) Infiltration for Perioperative Analgesia in Lumbosacral Spine Surgery: a Monocentric Randomized Trial.
Brief Title: Bilateral Erector Spinae Plane Block Versus Local Anesthetic Infiltration for Perioperative Analgesia in Spine Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Prof. Marco Rossi (Unknown); Dr. Roberta Nestorini (Unknown); Dr. Mariangela Di Muro (Unknown)
Responsible Party: Principal Investigator, VERGARI ALESSANDRO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP01
Record Dates: First submitted 2019-09-21; First posted 2019-10-10 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; SPINAL Fracture; Spondylolisthesis
Keywords: Analgesia, Patient-Controlled; Anesthetics, Local; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Spinal Fractures; Spondylolisthesis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block (Experimental): Ultrasound-guided, performed below erector spinae plane (ropivacaine 0.5% 20 mL each side).
  Interventions: Procedure: ESP block
- Wound infiltration (Active Comparator): Ropivacaine 0.5% 20-40 mL, performed by surgeon.
  Interventions: Procedure: Wound infiltration

INTERVENTIONS:
Procedure: ESP block — ESP block bilaterally performed at the level of the surgical site prior to surgery.
  Arms: ESP block
Procedure: Wound infiltration — Wound infiltration performed at the surgical site at the end of surgery.
  Arms: Wound infiltration

SUMMARY:
Postoperative pain still represents an important perioperative issue, affecting more than 80% of patients undergoing surgery. A suboptimal pain management doesn't just affects quality of life, but can compromise rehabilitation plan, increase morbidity and determine the development of chronic pain. Last but not least, far from being just an obligation for physicians, a good analgesia is a fundamental right of every patient.

In order to meet these important demands, a great number of guidelines has been provided, all of these underlying that the centerpiece of postoperative analgesia lies in the multimodality management, thereby combining different medications and different ways of delivering them, with the aim of targeting distinct receptor systems and improving efficacy, while limiting side effects.

In 2018, the investigators conducted a case-series analysis on 17 patients undergoing lumbar surgery to find out the role of Sublingual Sufentanil Tablet System (SSTS) in a multimodal analgesia regimen. Patients expressed a good pain relief, with most benefit during physiotherapy sessions and early discharges, in absence of side effects. Since then, SSTS has been part of regular clinical practice in our hospital.

The aim of this randomized trial is to examine the analgesic efficacy and the opioid sparing role in spine surgery of a recently developed regional anesthesia technique, the Erector Spinae Plane block (ESP block), as opposed to Local Anaesthetic (LA) wound infiltration.

The latter is a widespread, simple and unexpensive mean of providing postoperative analgesia. On the other hand, ESP block is an ultrasound-guided interfascial plain block, in which LA is injected below the erector spine muscle, closer to costotransverse foramina and origin of dorsal and ventral rami. It does provide an efficient multidermatomal sensory blockade (according to craniocaudal LA spread), with the advantage of being simple and safe.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for lumbar fusion surgery on account of vertebral fractures or degenerative spondylolisthesis.
* Patients consent.

Exclusion Criteria:

* Opioid tolerance;
* Documented sleep apnoea or home oxygen therapy;
* History of alcohol or drug abuse;
* Patients with an allergy or hypersensitivity to opioids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) at Post-Anesthesia Care Unit (PACU) arrival | At the end of surgery, at PACU arrival.
  NRS scale is a 11-point scale (0-11), with which patients self-report and rate level of breakthrough pain, where 0 is no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Difference in Pain Intensity Difference (PID) at PACU arrival, at 15 minutes, 30 minutes, 60 minutes, 2 hours, 6 hours from PACU arrival. | At the end of surgery, at PACU arrival; at 15 minutes, 30 minutes, 60 minutes, 2 hours, 6 hours from PACU arrival
  PID summarizes treatment response over a clinically relevant period. It represents a raw difference in pain intensity (i.e. the difference between the NRS value at each time point from the NRS at PACU arrival) and it is based on NRS data. It ranges from 0 to 10. The higher the value, the better the pain relief, since the greater is the pain intensity difference.
Difference in Sum of Pain Intensity Difference (SPID) at 12, 24, 48, 72 hours from PACU arrival. | 12 hours, 24 hours, 48 hours, 72 hours from PACU arrival.
  SPID is calculated multiplying the PID score at each time point by the duration (in hours) since the preceding time point, and then summing the values over the relevant time period. SPID represents the sum of the absolute difference in pain intensity. It ranges from 0 to an undefined value, variable according to the time weighted sum. The higher the value, the better the pain relief, since the greater is the pain intensity difference.
Number of Sublingual Sufentanil Tablets taken | 24 hours, 48 hours, 72 hours from PACU arrival.
  All patients eligible will be provided with Sufentanil Sublingual Tablet System.
Safety profile (incidence of adverse events) | Anytime during the study.
  Report of any adverse effect (sickness, vomiting, itching, numbness, respiratory side effects, procedure-related complications,..)
Patients satisfaction | Before discharge, an average of 48 hours from the end of surgery.
  All patients will fill out an Ease-Of-Care (EOC) Questionnaire, highlighting satisfaction with level of pain control and satisfaction with method of administration of pain medication.
Length of hospital stay | At discharge, an average of 48 hours from the end of surgery.
  Length of hospital stay after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico A. Gemelli, Rome, Italy